CLINICAL TRIAL: NCT04144101
Title: Comparison of Lower Dosage of Etoricoxib Versus Aceclofenac in the Treatment of Patients With Rheumatoid Arthritis: A Single-center, Parallel-group, Randomized Controlled Pilot Study
Brief Title: Etoricoxib vs Aceclofenac in the Treatment of Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Cheng-Chung Wei, Professor, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CS07005
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Rheumatoid Arthritis
Keywords: etoricoxib aceclofenac efficacy safety Taiwanese
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etoricoxib; aceclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Etoricoxib (Experimental): Etoricoxib 60 mg QD
  Interventions: Drug: Etoricoxib
- Aceclofenac (Experimental): Aceclofenac 100 mg BID
  Interventions: Drug: Aceclofenac

INTERVENTIONS:
Drug: Etoricoxib — Etoricoxib 60 mg QD Oral
  Other Names: Arcoxia
  Arms: Etoricoxib
Drug: Aceclofenac — Aceclofenac 100 mg BID Oral
  Other Names: TONEC
  Arms: Aceclofenac

SUMMARY:
Comparison of lower dosage etoricoxib (60 mg daily) with aceclofenac (100 mg bid) for their efficacy and safety in the treatment of rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
This was a single medical center, parallel-group, randomized controlled trial, which conducted for eight weeks. In this study, 40 patients of RA were randomly assigned to two different treatment groups (etoricoxib and aceclofenac), and 20 patients were enrolled for each group. In addition to baseline data collection, objective assessment tools were used to evaluate for efficacy and safety. The primary endpoint was American College of Rheumatology 20% improvement criteria (ACR20) , secondary endpoints were the ACR 50,70, disease activity score 28 (DAS 28), European League Against Rheumatism (EULAR) response criteria, the number of tender and swollen joints, physician's global assessment, patient's global assessment, pain scores, the short form health survey (SF-36) health Questionnaire and etc. In addition, all adverse reactions were recorded and all the results were analyzed in the intention to treat (ITT) manner.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis as Rheumatoid Arthritis

Exclusion Criteria:

* 1. Pregnant or breast-feeding women. 2. Chemotherapy or radiation therapy in cancer patients

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-03-01 (Actual); Primary Completion 2007-07-31 (Actual); Study Completion 2007-07-31 (Actual)

PRIMARY OUTCOMES:
American College of Rheumatology 20% improvement criteria (ACR20) | week 0, week 8
  The investigators use ACR20 to compared the difference between the week 8 and week 0

SECONDARY OUTCOMES:
American College of Rheumatology 50% improvement criteria (ACR50) | week 0, week 8
  The investigators use ACR50 to compared the difference between the week 8 and week 0
American College of Rheumatology 70% improvement criteria (ACR70) | week 0, week 8
  The investigators use ACR70 to compared the difference between the week 8 and week 0
Disease activity score 28 (DAS28) | week 0, week 8
  The investigators use DAS28 to compared the difference between the week 8 and week 0
European League Against Rheumatism (EULAR) response criteria | week 0, week 8
  The investigators use EULAR responder rate to compared the difference between the week 8 and week 0
The number of tender and swollen joints | week 0, week 8
  The investigators use the number of tender and swollen joints to compared the difference between the week 8 and week 0
Physician's global assessment (PhGA) | week 0, week 8
  The investigators use PhGA to compared the difference between the week 8 and week 0
Patient's global assessment (PGA) | week 0, week 8
  The investigators use PGA to compared the difference between the week 8 and week 0
Visual Analog Scale for pain (VAS) | week 0, week 8
  The investigators use VAS to compared the difference between the week 8 and week 0
Quality of life by SF-36 | week 0, week 8
  The investigators use SF-36 to compared the difference between the week 8 and week 0

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Ching Wei, Ph. D., Study Director — Chung Shan Medical University

IPD SHARING:
Plan to Share IPD: No